CLINICAL TRIAL: NCT01697969
Title: Confocal Analysis of Corneal Structures of Symptomatic Allergic Conjunctivitis Patients Pre and Post Treatment With Olopatadine HCL Ophthalmic Solution, 0.2%
Brief Title: Confocal Analysis of Corneal Structures of Symptomatic Allergic Conjunctivitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: M-12-047
Record Dates: First submitted 2012-09-27; First posted 2012-10-02 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-07

CONDITIONS: Allergic Conjunctivitis
Keywords: allergic conjunctivitis; Pataday; Olopatadine
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pataday (Experimental): Olopatadine hydrochloride ophthalmic solution, 0.2%, 1 drop once daily in both eyes for 14 days
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.2%

INTERVENTIONS:
Drug: Olopatadine hydrochloride ophthalmic solution, 0.2%
  Other Names: PATADAY®

SUMMARY:
The purpose of this study is to descriptively evaluate the corneal structures of allergic conjunctivitis patients.

DETAILED DESCRIPTION:
Heidelberg Retina Tomograph (HRT) will be used to descriptively evaluate the corneal structures and assess the immune cell status of allergic conjunctivitis patients pre- and post-treatment with olopatadine 0.2% in relation to a normative database.

ELIGIBILITY:
Inclusion Criteria:

* Read, sign, and date an Ethics Committee reviewed and approved informed consent form.
* Females of childbearing potential who:

  * Are not breast-feeding;
  * Do not intend to become pregnant for the duration of the study;
  * Are using adequate birth control methods and agree to continue for the duration of the study.
* Able to read, understand and answer questions by investigator.
* Willing and able to attend all required study visits and follow directions as stipulated by the protocol and investigator.
* History of allergic conjunctivitis (within the past 12 months) and active signs and symptoms of ocular allergies for which treatment is necessary, in the opinion of the investigator.
* Visual acuity correctable to 20/30 (Snellen) or better in each eye at distance with or without glasses correction.
* Ocular health within normal limits as determined by the investigator.
* No contact lens wear 14 days prior to enrollment and willing to not wear contact lenses for the duration of the study.
* Willing to follow a 14-day washout period due to contraindicated medication use, if deemed necessary by investigator.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Contraindications or hypersensitivity to the use of the test article or its components.
* Inability or unwillingness to follow all study instructions and complete study visits as required.
* Only one sighted eye or visual acuity not correctable to 20/30 (Snellen) in both eyes at the Screening Visit.
* Ocular trauma within 6 months prior to Visit 1 in either eye.
* Any ocular surgical intervention within six months prior to Visit 1 or anticipation of ocular surgery during the study.
* Presumed or actual ocular infection within 30 days prior to Visit 1.
* Any severe or serious ocular condition or significant illness.
* Any abnormal slit-lamp findings at the time of the Screening Visit.
* Contact lens wear within 14 days prior to the study start and unwillingness to undergo a wash-out period of 14 days; unwilling to not wear contact lenses for the duration of the study.
* Use of over-the-counter (OTC) ocular medications within the past 14 days unless willing to follow wash out period.
* Use of topical or systemic ocular medications requiring longer than a two-week washout period.
* Participation in any other investigational study in the 30-day period before entry into this study (i.e., Visit 1) or concomitantly with this study.
* Women who are pregnant, nursing, or of childbearing potential not utilizing adequate birth control measures.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Sindt, OD, FAAO, Principal Investigator — University of Iowa; Pam Kaur, MS PhD, Study Director — Alcon Research
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 1 study center located in the United States.
Pre-assignment Details: Of the 17 participants enrolled, 4 were exited from the study as screen failures prior to exposure to the test product. This reporting group includes all participants exposed to the test product (13).
Groups:
- Overall Study: Olopatadine hydrochloride ophthalmic solution, 0.2%, 1 drop once daily in both eyes for 14 days
Period: Overall Study
Arm/Group | Overall Study
Started | 13
Completed | 10
Not Completed | 3
Not completed — Did not meet inc/exc criteria | 3

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants exposed to the test product.
Arm/Group | Overall Study
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Patient-Assessed Ocular Itching
Description: The patient rated the severity of ocular itching using a predetermined 0-4 scale, where 0=none and 4=severe itching with irresistible urge to rub. Each eye was rated separately. A 2-week washout period from prior allergy medication (if applicable) preceded the baseline assessment.
Time Frame: Baseline (Day 1), Day 14
Population: The analysis population includes all participants exposed to the test product. Here, "n" is the number of participants with non-missing values at the specific time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Left Eye; Right Eye: Olopatadine hydrochloride ophthalmic solution, 0.2%, 1 drop once daily for 14 days
Arm/Group | Left Eye | Right Eye
Number analyzed (Participants) | 13 | 13
units on a scale
  Baseline (Day 1) | 2.2 (0.85) | 2.2 (0.92)
  Day 14 (n=11) | 0.5 (0.52) | 0.5 (0.52)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (October 11, 2012 to July 25, 2013). This analysis group includes all participants exposed to the test product.
Description: At each visit, after the subject had the opportunity to spontaneously mention any problems, the investigator inquired about AEs by asking the standard questions, "Have you had any health problems since your last study visit? Have there been any changes in the medicines you take since your last study visit?"
Arm/Group | Overall Study
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=13)
Arthropod infestation (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
The lack of concurrent control made it difficult to discriminate changes caused by PATADAY® from that caused by other factors, such as observer or patient expectation. Open-labeled design increased the bias from the observer or patient expectation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.